CLINICAL TRIAL: NCT04042246
Title: Knowledge on Vaccination Schedule and Full Immunization, and Its Effect on Vaccine Take-up in Jada Local Government Area in Adamawa State, Northeastern Nigeria
Brief Title: Effect of Knowledge on Vaccine Take-up in Adamawa State, Northeastern Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Ryoko Sato, Principal Investigator, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: TBDNA
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Immunization; Infection; Educational Problems; Information Seeking Behavior
MeSH Terms: conditions — Infections; Information Seeking Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention is implemented among Control
- Treatment (Educational Information on Vaccination) (Experimental): Provide general and tailored information on vaccination and vaccination schedule at the end of the baseline survey
  Interventions: Behavioral: Information Provision

INTERVENTIONS:
Behavioral: Information Provision — Provide the information on the importance of the vaccination and tailored vaccination schedule
  Arms: Treatment (Educational Information on Vaccination)

SUMMARY:
Child immunization is not a one-time behavior; rather, it is a repeated behavior within a specific timeframe. Not only the low immunization, but also the dropout of immunization and the delayed immunization from the recommended immunization schedule are prevalent and high in Africa. The most common reason for the incomplete vaccination is that caregivers thought the children had already been fully immunized (44.8%), according to Nigeria Multiple Indicator Cluster Survey (MICS) conducted in 2016/2017.

Caregivers' misconception of the complete immunization can be attributed to the complicated immunization schedule. In Nigeria, infants are supposed to receive 9 different types of vaccines at 5 different times within the first year since the births. To make things more complicated, the vaccine schedule changes over time; for example in Nigeria, the new vaccine, inactivated polio vaccine (IPV) was introduced in 2015 to be received at 14 weeks after births, and rotavirus vaccine and meningococcal A vaccine are scheduled for the introduction in 2019.

In this complicated and rapidly-changing environment regarding vaccination schedule, the goal of the study is to improve the understanding of vaccination completion and children's vaccination status among caregivers, which can then lead to the improved rate of full vaccination among children.

Objectives The main objectives of this study are to understand the impact of providing the general and tailored information on the vaccination schedule and vaccination status of women's children on the vaccine take-up. In this study, the investigators focus on women who has a child who is 12 months old or younger.

Hypothesis

The main hypothesis of this proposed study are as follows:

1. Information on vaccination among caregivers: the general and tailored information on vaccination schedule and child's vaccination status, improves the knowledge on benefit and understanding of vaccination completion, vaccination schedule and the vaccination status of the children among caregivers
2. Full immunization rate: through the improved knowledge level on the concept of vaccination completion and their children's vaccination status, the proposed study increases the full immunization rate among children

DETAILED DESCRIPTION:
Background and Objectives Despite the proven benefit of vaccines, the child immunization rate has been stagnant and the rate in African countries lags behind other regions in the world. For example, the global coverage of three doses diphtheria-tetanus-pertussis (DPT3) has been stagnant at 85% since 2015, while DPT3 coverage in Africa remains at 72% since 2010. The distribution of unvaccinated children is unequal; out of about 20 million infants who are not fully vaccinated, more than 20 percent of them reside in three countries, including Nigeria, the proposed study site. Furthermore, Nigeria is one of the few countries where the coverage of DPT3 coverage has decreased over time: 54 percent in 2010 to 42 percent in 2017.

Child immunization is not a one-time behavior; rather, it is a repeated behavior within a specific timeframe. Not only the low immunization, but also the dropout of immunization and the delayed immunization from the recommended immunization schedule are prevalent and high in Africa. The most common reason for the incomplete vaccination is that caregivers thought the children had already been fully immunized (44.8%), according to Nigeria Multiple Indicator Cluster Survey (MICS) conducted in 2016/2017.

Caregivers' misconception of the complete immunization can be attributed to the complicated immunization schedule. Each type and dose of vaccine has its own significance in terms of the type of preventable disease and the achievable efficacy level. In Nigeria, infants are supposed to receive 9 different types of vaccines at 5 different times within the first year since the births. For example, oral poliovirus vaccine (OPV) is to protect infants from contracting polio, a highly contagious disease. At present, Nigeria is one of the three countries in the world, which have not eliminated polio. Infants are scheduled to receive OPV four times; at birth, 6, 10, and 14 weeks. The efficacy of the first dose OPV (oral polio vaccine) is 82%, while the second and the third doses are 90% and 99% or more, respectively. To make things more complicated, the vaccine schedule changes over time; for example in Nigeria, the new vaccine, inactivated polio vaccine (IPV) was introduced in 2015 to be received at 14 weeks after births, and rotavirus vaccine and meningococcal A vaccine are scheduled for the introduction in 2019.

In this complicated and rapidly-changing environment regarding vaccination schedule, the goal of the study is to improve the understanding of vaccination completion and children's vaccination status among caregivers, which can then lead to the improved rate of full vaccination among children.

Objectives The main objectives of this study are to understand the impact of providing the general and tailored information on the vaccination schedule and vaccination status of women's children on the vaccine take-up. This study focuses on women who has a child who is 12 months old or younger.

Hypothesis

The main hypothesis of this proposed study are as follows:

1. Information on vaccination among caregivers: the general and tailored information on vaccination schedule and child's vaccination status, improves the knowledge on benefit and understanding of vaccination completion, vaccination schedule and the vaccination status of the children among caregivers
2. Full immunization rate: through the improved knowledge level on the concept of vaccination completion and their children's vaccination status, the proposed study increases the full immunization rate among children

Literature Review Knowledge is powerful in shaping people's health behaviors. In a situation where the health behaviors among the population do not reach the optimal level, one obvious way to attempt to improve the situation is to provide the information to encourage the population for adopting the health behaviors.

In case of vaccination, information provision has a great potential to increase the take-up of vaccination, especially in places where one of the main perceived barriers is the lack of knowledge on the vaccination schedule, as is the case in Adamawa state.

However, the effectiveness of information provision on the vaccine take-up might differ, depending on the type of information provided. One study provided the information on the benefit of tetanus vaccines to caregivers in India and they found the strong effect of the information provision on the vaccine take-up. The effectiveness of gain-framed and loss-framed messaging was statistically identical in their study. On the other hand, salient information, such as fear appeals, might be ineffective or it can even backfire. The investigators found, in the previous project, that in Jada Local Government Area, fear appeals intervention backfired on the tetanus-toxoid vaccine take-up among women who never received the vaccine.

If caregivers are not aware of the vaccination schedule as found in MICS 2016/2017, simply providing the information on the next vaccination schedule can be effective. Recent technological advancement makes it easy and cost-effective to send the reminder through SMS message.

Although SMS (Short Message Service) reminders are found to be effective in affecting one-time vaccine take-up, this intervention should be accompanied with the provision of more fundamental information, which can induce the repeated vaccination behaviors, to make the effect of intervention sustainable. This study proposes to provide fundamental information, which informs respondents the overall vaccination schedule, as well as tailored information, which informs where their children are in the vaccination schedule. The investigators hypothesize that, once respondents understand the overall vaccination schedule, it is easy to comprehend when and how many times more they should visit the clinic, instead of fully relying on the supply-side intervention such as SMS reminders.

ELIGIBILITY:
Inclusion Criteria:

* women with a child 12 months old or younger

Exclusion Criteria:

* exclude women who do not have a child 12 months or younger

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-02-09 (Actual)

PRIMARY OUTCOMES:
Number of participants who have the accurate knowledge level of vaccination, as assessed by survey questionnaire | 2 weeks
  The investigators will collect the information on respondents' knowledge on vaccination through surveys. The knowledge level is calculated from 5 questions: 1) the number of type of vaccines a child needs to receive before 12 months old, 2) the number of times a child needs to receive Pentavalent vaccine, 3) the last month when a child needs to receive Pentavalent vaccine, 4) the timing when a child needs to receive BCG vaccine, and 5) the number of clinic visits (at minimum) a child needs to make for complete vaccination. For each question, the score is 0 if wrong, or 1 if correct.
  The knowledge level scale ranges from 0 to 5, which is the total number of correct answers.
Number of participants who bring their children for the full vaccination, as assessed by the follow-up tracking survey at health clinics | 9 months
  The investigators will collect the information on the actual vaccination status among respondents' children

CONTACTS AND LOCATIONS:
Overall Officials: Ryoko Sato, Ph.D., Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Jada Local Government Primary Health Care Development Agency, Jada, Adamawa, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bolu O, Nnadi C, Damisa E, Braka F, Siddique A, Archer WR, Bammeke P, Banda R, Higgins J, Edukugo A, Nganda GW, Forbi JC, Liu H, Gidado S, Soghaier M, Franka R, Waziri N, Burns CC, Vertefeuille J, Wiesen E, Adamu U. Progress Toward Poliomyelitis Eradication - Nigeria, January-December 2017. MMWR Morb Mortal Wkly Rep. 2018 Mar 2;67(8):253-256. doi: 10.15585/mmwr.mm6708a5. PMID 29494568
- [Background] Feldstein LR, Mariat S, Gacic-Dobo M, Diallo MS, Conklin LM, Wallace AS. Global Routine Vaccination Coverage, 2016. MMWR Morb Mortal Wkly Rep. 2017 Nov 17;66(45):1252-1255. doi: 10.15585/mmwr.mm6645a3. PMID 29145357
- [Background] Kazungu JS, Adetifa IMO. Crude childhood vaccination coverage in West Africa: Trends and predictors of completeness. Wellcome Open Res. 2017 Feb 15;2:12. doi: 10.12688/wellcomeopenres.10690.1. PMID 28459105
- [Background] Kim-Farley RJ, Rutherford G, Lichfield P, Hsu ST, Orenstein WA, Schonberger LB, Bart KJ, Lui KJ, Lin CC. Outbreak of paralytic poliomyelitis, Taiwan. Lancet. 1984 Dec 8;2(8415):1322-4. doi: 10.1016/s0140-6736(84)90831-6. PMID 6150332
- [Background] Lukusa LA, Ndze VN, Mbeye NM, Wiysonge CS. A systematic review and meta-analysis of the effects of educating parents on the benefits and schedules of childhood vaccinations in low and middle-income countries. Hum Vaccin Immunother. 2018;14(8):2058-2068. doi: 10.1080/21645515.2018.1457931. Epub 2018 May 14. PMID 29580159
- [Background] Manakongtreecheep K. SMS-reminder for vaccination in Africa: research from published, unpublished and grey literature. Pan Afr Med J. 2017 Jun 22;27(Suppl 3):23. doi: 10.11604/pamj.supp.2017.27.3.12115. eCollection 2017. PMID 29296158
- [Background] Mbengue MAS, Mboup A, Ly ID, Faye A, Camara FBN, Thiam M, Ndiaye BP, Dieye TN, Mboup S. Vaccination coverage and immunization timeliness among children aged 12-23 months in Senegal: a Kaplan-Meier and Cox regression analysis approach. Pan Afr Med J. 2017 Jun 21;27(Suppl 3):8. doi: 10.11604/pamj.supp.2017.27.3.11534. eCollection 2017. PMID 29296143
- [Background] Mutua MK, Kimani-Murage E, Ngomi N, Ravn H, Mwaniki P, Echoka E. Fully immunized child: coverage, timing and sequencing of routine immunization in an urban poor settlement in Nairobi, Kenya. Trop Med Health. 2016 May 16;44:13. doi: 10.1186/s41182-016-0013-x. eCollection 2016. PMID 27433132
- [Background] Powell-Jackson T, Fabbri C, Dutt V, Tougher S, Singh K. Effect and cost-effectiveness of educating mothers about childhood DPT vaccination on immunisation uptake, knowledge, and perceptions in Uttar Pradesh, India: A randomised controlled trial. PLoS Med. 2018 Mar 6;15(3):e1002519. doi: 10.1371/journal.pmed.1002519. eCollection 2018 Mar. PMID 29509769
- [Background] Tannenbaum MB, Hepler J, Zimmerman RS, Saul L, Jacobs S, Wilson K, Albarracin D. Appealing to fear: A meta-analysis of fear appeal effectiveness and theories. Psychol Bull. 2015 Nov;141(6):1178-204. doi: 10.1037/a0039729. PMID 26501228
- [Background] VanderEnde K, Gacic-Dobo M, Diallo MS, Conklin LM, Wallace AS. Global Routine Vaccination Coverage - 2017. MMWR Morb Mortal Wkly Rep. 2018 Nov 16;67(45):1261-1264. doi: 10.15585/mmwr.mm6745a2. PMID 30439873
- [Background] Jacobson Vann JC, Jacobson RM, Coyne-Beasley T, Asafu-Adjei JK, Szilagyi PG. Patient reminder and recall interventions to improve immunization rates. Cochrane Database Syst Rev. 2018 Jan 18;1(1):CD003941. doi: 10.1002/14651858.CD003941.pub3. PMID 29342498